CLINICAL TRIAL: NCT04940117
Title: Improve eGFR in Chronic Kidney Disease
Brief Title: Effects of the Eefooton on eGFR and QoL in Chronic Kidney Disease Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Jin-Shuen Chen, Chair of IRB, Kaohsiung Veterans General Hospital.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB No. KSVGH21-CT5-19
Record Dates: First submitted 2021-06-22; First posted 2021-06-25 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Chronic Kidney Diseases
Keywords: eGFR
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Chronic Kidney Disease before dialysis
Masking Description: Patients with renal failure with Eefooton oral solution for six months and blood test to check the changes in eGFR values
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- blood test data before and after taking (Experimental): Checking eGRF value before and after taking Eefooton oral solution
  Interventions: Dietary Supplement: Eefooton oral solution

INTERVENTIONS:
Dietary Supplement: Eefooton oral solution — Check eGFR value, liver and kidney function every month

SUMMARY:
Chronic renal failure is a chronic and progressive disease with a poor prognosis. In recent years, it can be found in many literature reports that traditional Chinese medicine therapy has obvious effects on early and mid-term chronic renal failure. It can not only improve clinical symptoms, but also block or delay the process of renal failure. It is relatively rare that compounds such as compounds. The side effects of drugs may be used in combination with compound drugs to improve clinical side effects and help patients improve their quality of life to complete the treatment course. It can provide clinicians with another choice in treatment. A previous study confirmed that the use of Eefooton oral solution of Chinese herbal medicine concentrate has a significant protective effect on the kidneys that have not undergone hemodialysis. Eefooton is extracted from Rhodiola, Huang Qi, American Ginseng, Dang Ginseng, and Ligustrum lucidum by biotechnology. It has immunomodulatory effects, anti-oxidation and anti-inflammatory effects, and regulates calcium metabolism. The purpose of this clinical observation and research is to evaluate the eGFR changes in the renal function of patients with chronic kidney disease with the combination of Eefooton oral solution and commonly used chemical drugs.

DETAILED DESCRIPTION:
The Blood test items consisted Blood urea nitrogen (BUN), Serum creatinine (SCr), estimated glomerular filtration rate (eGFR), serum Uric acid, plasma Albumin (ALB), Hemoglobin (Hb), Alkaline phosphatase (ALP), Serum Glutamic-Oxalocetic Transaminase (SGOT), Serum glutamic pyruvic transaminase (SGPT), Glucose(AC), Serum sodium, Serum potassium, Corrected calcium , Phosphorus (Blood). Glycated hemoglobin (HbA1c), Triglyceride (TG), Total cholesterol (Chol), High-density lipoprotein (HDL), Low-density lipoprotein (LDL). During the entire research process did not change diet, lifestyle, habits and the use of drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic kidney disease who have signed the subject's consent and the glomerular filtration rate (eGFR) is less than 59ml/min/1.73m2
2. Both male and female patients aged 20-85 years old are acceptable
3. You must be able to come back at a specific time each month during the 6-month trial

Exclusion Criteria:

If you have any of the following conditions, you will not be able to participate in this research project:

1. Drug abuse.
2. Heart failure (stage 3-4)
3. Mental illness (psychotic disorder, epilepsy, depression, panic disorder)
4. Patients who have undergone dialysis or are expected to have a kidney transplant in the last three months
5. The blood pressure still exceeds 150/90mmHg after using more than three antihypertensive drugs
6. Pregnancy or planning to become pregnant or breastfeeding
7. Malignant disease
8. Acute illness (hepatitis, jaundice, acute myocardial infarction) in the last 3 months
9. The patient is engaged in another research study.
10. 3 months before entering the study or having used NSAIDs, anti-rejection drugs or performing imaging agent examinations during the study
11. You have participated in other research study in the previous month
12. You have drug dependence and drinking habits

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
QoL | one months
  The SF-36 questionnaire as assessment of the safety that consists physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality (fatigue), social functioning, role limitations due to emotional health, and general mental health.

OTHER OUTCOMES:
eGFR | one months
  The eGFR value is an important marker for kidney function. The GFR unit is ml/min/1.73m2

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Shuen Chen, Ph.D, Principal Investigator — Kaohsiung Veterans General Hospital.; Sam-Chiang Wu, Ph.D, Study Director — WU SAM-CHIANG Medical clinic
Locations (1):
- WU SAM-CHIANG Medical clinic, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No